CLINICAL TRIAL: NCT06264271
Title: The Effect of Nutrition Education on Glycemic Control in Patients With Type 1 Diabetes Initiating the Use of Glucose Sensors
Brief Title: The Effect of Nutrition Education on Glycemic Control in Patients With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Eva Horová, MD, Principal Investigator, Charles University, Czech Republic
Other Study IDs: GIP-22-NL-06-203
Record Dates: First submitted 2024-02-12; First posted 2024-02-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: carbohydrate counting; flexible insulin dosing; structured education; glycemic control; glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with nutrition education: Patients who experienced at least one structured education session between 24 months before sensor initiation and 6 months after sensor initiation were allocated to the group with education.
  Interventions: Behavioral: structured nutrition intervention
- Group without nutrition education: Patients who received standard care, which may have included short education during routine visits or self-education through online resources or educational materials, were assigned into the group without education.

INTERVENTIONS:
Behavioral: structured nutrition intervention — Structured nutrition education on carbohydrate counting and flexible insulin dosing by qualified nutritionist.
  Groups: Group with nutrition education

SUMMARY:
The study aims to elucidate whether patients with T1D initiating sensor monitoring experience greater improvement in glycemic control (HbA1c) when provided with structured nutrition education compared to those initiating sensor monitoring without such education.

DETAILED DESCRIPTION:
Education on carbohydrate counting and flexible insulin dosing improves glycemic control, which is also enhanced by glucose sensor usage. However, the combined effect of structured education and the initiation of sensor monitoring remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* type 1 diabetes duration for at least 12 months prior to sensor initiation
* glucose sensor monitoring initiated at the Diabetes Centre of the General University Hospital in Prague

Exclusion Criteria:

* uncertain diabetes type
* pregnancy
* change or suspension of glucose sensor monitoring during the study period
* unavailability of sensor data
* automated insulin delivery treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age ≥ 18 years, T1D duration for at least 12 months prior to sensor initiation, and all sensor monitoring initiated at the Diabetes Centre of the General University Hospital in Prague.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
difference in HbA1c | at month 12
  the difference in HbA1c between the groups with and without education

SECONDARY OUTCOMES:
differences in time in range | at month 12
  differences in time in range (percentages) (70-180 mg/dL [3.9-10.0 mmol/L]) between groups with and without education
differences in time below range | at month 12
  differences in time below range (percentages) in level 1 hypoglycemia (54-69 mg/dL [3.0-3.8 mmol/L]), level 2 hypoglycemia (<54 mg/dL [<3.0 mmol/L]) between groups with and without education
differences in time above range | at month 12
  differences in time above range (percentages) (>181 mg/dL [>10.1 mmol/L]) between groups with and without education
differences in coefficient of variation | at month 12
  differences in coefficient of variation between groups with and without education

CONTACTS AND LOCATIONS:
Overall Officials: Eva Horová, Principal Investigator — 3rd Department of Internal Medicine, 1st Faculty of Medicine, Charles University, Prague, Czechia
Locations (1):
- Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DAFNE Study Group. Training in flexible, intensive insulin management to enable dietary freedom in people with type 1 diabetes: dose adjustment for normal eating (DAFNE) randomised controlled trial. BMJ. 2002 Oct 5;325(7367):746. doi: 10.1136/bmj.325.7367.746. PMID 12364302
- [Background] Shearer A, Bagust A, Sanderson D, Heller S, Roberts S. Cost-effectiveness of flexible intensive insulin management to enable dietary freedom in people with Type 1 diabetes in the UK. Diabet Med. 2004 May;21(5):460-7. doi: 10.1111/j.1464-5491.2004.01183.x. PMID 15089791
- [Background] Elbalshy M, Haszard J, Smith H, Kuroko S, Galland B, Oliver N, Shah V, de Bock MI, Wheeler BJ. Effect of divergent continuous glucose monitoring technologies on glycaemic control in type 1 diabetes mellitus: A systematic review and meta-analysis of randomised controlled trials. Diabet Med. 2022 Aug;39(8):e14854. doi: 10.1111/dme.14854. Epub 2022 Apr 25. PMID 35441743
- [Background] Maiorino MI, Signoriello S, Maio A, Chiodini P, Bellastella G, Scappaticcio L, Longo M, Giugliano D, Esposito K. Effects of Continuous Glucose Monitoring on Metrics of Glycemic Control in Diabetes: A Systematic Review With Meta-analysis of Randomized Controlled Trials. Diabetes Care. 2020 May;43(5):1146-1156. doi: 10.2337/dc19-1459. PMID 32312858
- [Background] Vigersky RA. The benefits, limitations, and cost-effectiveness of advanced technologies in the management of patients with diabetes mellitus. J Diabetes Sci Technol. 2015 Mar;9(2):320-30. doi: 10.1177/1932296814565661. PMID 25555391
- [Derived] Navratilova V, Zadakova E, Soupal J, Skrha J Jr, Do QD, Radovnicka L, Haskova A, Prazny M, Horova E. The Effect of Nutrition Education on Glycemic Outcomes in People With Type 1 Diabetes Initiating the Use of Glucose Sensors. Endocrinol Diabetes Metab. 2025 Mar;8(2):e70047. doi: 10.1002/edm2.70047. PMID 40121673